CLINICAL TRIAL: NCT00320437
Title: The Intergenerational Transmission of Trauma From Terror: A Developmental Perspective
Brief Title: Intergenerational Transmission of Terror
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: terror HMO-CTIL
Record Dates: First submitted 2006-04-30; First posted 2006-05-03 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-11

CONDITIONS: Anxiety; Trauma; Stress Disorders
Keywords: trauma; anxiety; antenatal; mothers; children; Gene x Environment Interaction
MeSH Terms: conditions — Anxiety Disorders; Wounds and Injuries; Stress Disorders, Traumatic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Our aim is examine avenues by which mothers can transmit their trauma to their children.

DETAILED DESCRIPTION:
The goal of the study is to test for genetic bases and Gene x Environment interactions on the development of difficulties, particularly stress disorders, in young children whose mother were exposed to terror before they were born.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were exposed to terror in the last 5 years
* Matched Controls

Exclusion Criteria:

* Does not speak Hebrew or English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-05; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Faraone, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Hadassah University Hospital, Jerusalem, Ein Kerem, Israel